CLINICAL TRIAL: NCT01984541
Title: Biological Standardization of Artemisia Vulgaris Allergen Extract to Determine the Biological Activity in Histamine Equivalent Units (HEP).
Brief Title: To Determine the Minimum Amount of Artemisia Vulgaris Allergen Extract Producing a Positive Skin Reaction.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laboratorios Leti, S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 6058-PR-PRI-200; 2013-001310-15 (EudraCT Number)
Record Dates: First submitted 2013-11-08; First posted 2013-11-14 (Estimated); Last update posted 2015-01-05 (Estimated); Status verified 2013-05

CONDITIONS: Allergy to Pollen
Keywords: Pollen
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Artemisia vulgaris allergen extract(four concentrations 10, 1, 0,1 y 0,01 mg/ml) Positive Control Negative Control
  Interventions: Biological: Artemisia vulgaris

INTERVENTIONS:
Biological: Artemisia vulgaris — Four concentrations of Artemisia vulgaris allergen extract, together with a positive and negative control will be tested in every patient in duplicate on the volar surface of the forearm.
  Other Names: Four different concentrations of Artemisia vulgaris allergen extract, positive control and negative control

SUMMARY:
The objective of this study is to determine the biological activity of Artemisia vulgaris allergen extract in histamine equivalent units (HEP) units, in order to be used as in-house reference preparation (IHRP).

DETAILED DESCRIPTION:
This is an open, unblinded and non-randomized biological assay. Tehe study design is a slight modification of the recommendations proposed by the Nordic Guidelines.

Four concentrations of Artemisia vulgaris allergen extract, together with a positive and negative control, using 10 mg/ml histamine dihydrochloride solution and a glycerinated phenol saline solution, respectively, will be tested in every patient in duplicate on the volar surface of the forearm.

ELIGIBILITY:
Inclusion Criteria:

Positive clinical history of inhalatory allergy to Artemisia vulgaris. Subject has provided written informed consent, appropriately signed and dated by the subject.

Subject can be male or female of any race and ethinic group. Age major or equal 18 years and ninor or equal 60 years at the study inclusion day.

A positive prick test with a standardized commercially Artemisia vulgaris allergen extract (Wheal medium diameter ≤ 3mm or wheal area ≥ 7 mm2). The skin prick test results are valid if performed within one year prior to the inclusion of the subject in the study.

A positive test for specific IgE to Artemisia vulgaris (CAP-RAST major or equal to 2). IgE results are valid if performed within one year prior to the inclusion of the subject in the study.

Allergy symptoms during the Artemisia vulgaris pollen season.

Exclusion Criteria:

Immunotherapy in the past 5 years with an allergen extract Artemisia vulgaris or other allergen extract that may interfere with the allergene to be tested (for example: Helianthus annuus (sunflower) elatior Ambrosia eiator (ambrosia) or peach.

Use of drugs that may interfere before and after with the skin reactions (for example: antihistamines).

Treatment with any of the following medications: oral tricyclic or tetracyclic antidepressants, beta-blockers, corticosteroids (major 10 mg/daily of prednisone or equivalent).

Women who are pregnant or breastfeeding period and women with positive pregnancy test at Visit 2, before skin prick test.

Dermographism affecting the skin area at the test site at either study visit. Atopic dermatitis affecting the skin area at the test site at either study visit. Urticaria affecting the skin area at the test site at either study visit. Diseases of the immune system relevant clinically, both autoimmune and immunodeficiencies.

Serious diseases not controlled that may increase the risk for the safety of the subjects involved in this study, including, but not limited to the following: heart failure, uncontrolled or severe respiratory diseases, endocrine diseases, clinically relevant kidney or liver diseases or hematological diseases. Participation in any other clinical trial within 30 days (or 5 times the biological half-life of the research of the study product, whichever is longer) prior to the inclusion of the subject in this clinical trial.

Patients with diseases or conditions that limit the use of adrenaline. Severe psychiatric, psychological or neurological disorders. Abuse of alcohol, drugs or medicines in the previous year. Subjects who have received anti-IgE (Omalizumab).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-03; Primary Completion 2014-06 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Wheal size area (mm2) on the skin at the site of the puncture during the immediate phase. | 15-20 min after aplication

CONTACTS AND LOCATIONS:
Overall Officials: Lena Erbiti, Study Chair — Laboratorios Leti, S.L.U
Locations (2):
- Spain (2):
  - Hospital de La Agencia Valenciana de Salud Vega Baja, Orihuela, Alicante
  - Hospital Clinic de Barcelona, Barcelona, Barcelona